CLINICAL TRIAL: NCT03396185
Title: Icotinib as Consolidation Therapy After Synchronous or Sequential Chemoradiotherapy in Stage IIIA-IIIB Non-small Cell Lung Cancer With EGFR Sensitive Mutation: A Single Center, Single Arm, Open Label and Prospective Clinical Study
Brief Title: Icotinib as Consolidation Therapy After Chemoradiotherapy in EGFR-Mutant Stage IIIA-IIIB Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-069
Record Dates: First submitted 2017-12-28; First posted 2018-01-10 (Actual); Last update posted 2018-07-18 (Actual); Status verified 2018-01

CONDITIONS: EGFR Gene Mutation; Non Small Cell Lung Cancer Stage IIIA; Non Small Cell Lung Cancer Stage IIIB
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Icotinib (Experimental): Patients with EGFR-mutant stage IIIA-IIIB and unresectable lung adenocarcinoma will receive Icotinib with a dose of 125 mg three times per day orally till progressive disease or unaccepted toxicity as consolidation therapy after synchronous or sequential chemoradiotherapy.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Patients who have EGFR-mutant stage IIIA-IIIB and unresectable lung adenocarcinoma will receive Icotinib with a dose of 125 mg three times per day orally till progressive disease or unaccepted toxicity as consolidation therapy after synchronous or sequential chemoradiotherapy.
  Other Names: Conmana

SUMMARY:
The main purpose of this study is to evaluate the relapse free survival of patients who have EGFR-mutant stage IIIA-IIIB Non-small Cell Lung Cancer and receive Icotinib as consolidation therapy after synchronous or sequential chemoradiotherapy.

DETAILED DESCRIPTION:
This is a single center, single arm, open label and prospective clinical study. Patients who have EGFR-mutant stage IIIA-IIIB and unresectable lung adenocarcinoma will receive Icotinib as consolidation therapy after synchronous or sequential chemoradiotherapy. The primary objective of this study is relapse free survival. The secondary objectives are overall survival, the frequency of adverse events and patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable stage IIIA-IIIB Non-small Cell Lung Cancer, histology or cytology confirmed lung adenocarcinoma, pathological specimens with EGFR 19 del and/or 21 L858R gene mutation detected by amplification refractory mutation system method
* Before receiving synchronous or sequential chemoradiotherapy, no metastasis detected by head MRI, bone scan, chest enhanced CT scan and the abdominal (including dual adrenal) enhanced CT scan
* Only received synchronous or sequential chemoradiotherapy as anti-tumor treatment; after that, chest enhanced CT showed no progressive disease (including Complete Response, Partial Response and Stable Disease )
* Platinum-based chemotherapy regimen, including: vinorelbine, docetaxel, paclitaxel, pemetrexed, etoposide, etc and combination of platinum (including but not limited to cisplatin and carboplatin)
* 3DCRT or IMRT radiotherapy technology with a dose of 95% PTV 60-66gy, 2Gy once daily, 5 times weekly, up to 30-33 times
* ECOG score 0-1
* Able to enter the group within 4-12 weeks after the completion of synchronous or sequential chemoradiotherapy
* Expected survival more than 12 weeks

Exclusion Criteria:

* Other malignant tumors within five years, except for completely cured cervical carcinoma, basal or squamous cell carcinoma
* In addition to synchronous or sequential chemoradiotherapy, ever received other systemic anti-tumor treatment, including chemotherapy or targeted therapy
* Any unstable systemic disease, including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, liver, kidney or metabolic disease
* Upper vena cava syndrome at baseline
* Idiopathic pulmonary fibrosis detected by CT at baseline
* Definite neurological or psychiatric disorders, including epilepsy or dementia
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Relapse Free Survival of participants | three years
  Relapse Free Survival was defined as the time from randomization to relapse of disease or death from any cause.

SECONDARY OUTCOMES:
Overall survival of participants | three years
  Overall survival was defined as the time from participants' randomization to their death due to any cause.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | three years
  The number of participants with treatment-related adverse events as assessed by CTCAE v4.0 would be recorded and calculated after them participating into the study and taking the experimental drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Science, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes